CLINICAL TRIAL: NCT05880134
Title: Cartilage Graft Reinforcement for Posterior Nasal Nerve Neurectomy in Allergic Rhinitis Surgeries; Randomized Controlled Trial.
Brief Title: Graft Reinforcement for Posterior Nasal Nerve Neurectomy in Allergic Rhinitis Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohammad Mahmoud Aouf, assistant lecturer, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MKSU 51-2-13
Record Dates: First submitted 2023-03-16; First posted 2023-05-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neurectomy
Keywords: allergic rhinitis; neurectomy; cartilage
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional posterior nerve neurectomy (Active Comparator): A vertical incision is made behind the posterior fontanelle. The posterior end of the posterior fontanelle is identified by palpation with an elevator. .
  The mucoperiosteum is raised gently using a Cottle elevator or a suction freer elevator, after making the initial incision. Care must be taken not to injure the sphenopalatine vessel during flap elevation.
  The peripheral part of the posterior nasal nerve can usually be identified just behind the incision, about 4-5 mm inferior to the sphenopalatine artery or crista ethmoidalis.
  I After identifying the nerve fibres, it is cauterised using monopolar suction cautery and cut using microscissors. It is essential to carry out this procedure on both sides for effective results.
  Interventions: Procedure: conventional posterior nerve neurectomy
- cartilage reinforcement after posterior nerve neurectomy (Active Comparator): A vertical incision is made behind the posterior fontanelle. The posterior end of the posterior fontanelle is identified by palpation with an elevator. .
  The mucoperiosteum is raised gently using a Cottle elevator or a suction freer elevator, after making the initial incision. Care must be taken not to injure the sphenopalatine vessel during flap elevation.
  The peripheral part of the posterior nasal nerve can usually be identified just behind the incision, about 4-5 mm inferior to the sphenopalatine artery or crista ethmoidalis.
  I After identifying the nerve fibres, it is cauterised using monopolar suction cautery and cut using microscissors. It is essential to carry out this procedure on both sides for effective results.
  Interventions: Procedure: cartilage graft reinforcement after posterior nerve neurectomy

INTERVENTIONS:
Procedure: conventional posterior nerve neurectomy — A vertical incision is made behind the posterior fontanelle. The posterior end of the posterior fontanelle is identified by palpation with an elevator. .
  The mucoperiosteum is raised gently using a Cottle elevator or a suction freer elevator, after making the initial incision. Care must be taken not to injure the sphenopalatine vessel during flap elevation.
  The peripheral part of the posterior nasal nerve can usually be identified just behind the incision, about 4-5 mm inferior to the sphenopalatine artery or crista ethmoidalis.
  I After identifying the nerve fibres, it is cauterised using monopolar suction cautery and cut using microscissors. It is essential to carry out this procedure on both sides for effective results.
  Arms: conventional posterior nerve neurectomy
Procedure: cartilage graft reinforcement after posterior nerve neurectomy — A vertical incision is made behind the posterior fontanelle. The posterior end of the posterior fontanelle is identified by palpation with an elevator. .
  The mucoperiosteum is raised gently using a Cottle elevator or a suction freer elevator, after making the initial incision. Care must be taken not to injure the sphenopalatine vessel during flap elevation.
  The peripheral part of the posterior nasal nerve can usually be identified just behind the incision, about 4-5 mm inferior to the sphenopalatine artery or crista ethmoidalis.
  I After identifying the nerve fibres, it is cauterised using monopolar suction cautery and cut using microscissors. It is essential to carry out this procedure on both sides for effective results.
  then harvest cartilage from nasal septum and refashion it around sphenopalatine bundle to prevent nerve re-innervation
  The mucoperiosteal flaps are repositioned . No nasal packing is required. Patients are discharged on the same day
  Arms: cartilage reinforcement after posterior nerve neurectomy

SUMMARY:
Rhinitis is defined clinically as having two or more symptoms of anterior or posterior rhinorrhea, sneezing, nasal blockage and/or itching of the nose during two or more consecutive days for more than 1 h on most days.

Allergic rhinitis is diagnosed when these symptoms are caused by allergen exposure leading to an IgE mediated reaction. The inflammatory mediators produced because of this IgE mediated reaction causes the classical symptoms of allergic rhinitis.

Nerve irritation causes sneezing and itching, the loss of mucosal integrity causes rhinorrhea, and the vascular engorgement leads to nasal blockage.

Based on the nasal symptoms the prevalence of allergic rhinitis in the Indian population is 20-30%.

Allergic rhinitis significantly affects the quality of life, it contributes to missed or unproductive time at school or work, disturbed sleep pattern and daytime somnolence.

The most popular and widely accepted treatment strategy for allergic rhinitis is pharmacotherapy, this includes antihistamines, leukotriene receptor antagonist and intranasal corticosteroids. These medical modalities are symptomatically effective in mild cases, with temporary relief and addressable adverse effects. Prolonged treatment with allergy immunotherapy causes a sustainable financial burden while remaining inaccessible at smaller towns.

Rhinorrhea is a frequent symptom reported amongst patients with allergic and vasomotor rhinitis. Most of these patients usually respond well to medical treatment.

Indications for surgical treatment are warranted only when medical treatment fails, or a patient wants a permanent solution.

In 1961, Golding-Wood first described vidian neurectomy for the treatment of allergic and vasomotor rhinitis. There was a high incidence of post-operative complications, such as disturbed lacrimal secretion and numbness of the cheek and gums. In 2007, Kikawada reported an endoscopic technique involving resection of the posterior nasal nerve near the sphenopalatine artery. With this technique, any intra-operative bleeding can be controlled under direct vision. In 2008, Ikeda et al. described submucosal reduction of the inferior turbinate and resection of the posterior nasal nerve. This resulted in significant improvements in nasal symptoms for patients with resistant chronic rhinitis (rhinorrhea).

The posterior nasal nerve is a peripheral branch of the sphenopalatine ganglion. It enters the nasal cavity through a separate foramen, 4-5 mm below the sphenopalatine foramen, after bifurcation of the nerve into the lacrimal nerve. The posterior superior nasal nerves innervate the superior and middle turbinates, and the superior and middle meatus.

Other parasympathetic nerve fibres of the nose branch off and joins the greater palatine nerve and enters the nasal cavity through the canaliculi in the perpendicular plate of the palatine bone as the posterior inferior nasal nerves. These nerves innervate the inferior turbinate and the inferior meatus.

DETAILED DESCRIPTION:
Allergic rhinitis (AR) is a growing health problem all over the world. Around the world, more than 500million subjects complained of AR, and its prevalence had been increased during the last decades . AR affected approximately 113 million people in Europe and about 30 - 60 million in the United States. Poorly controlled symptoms of AR could lead to different comorbidities (e.g., impaired sleep with consequent daytime fatigue which affect overall patient's work or school achievement; all affect quality of life (QoL) with increased treatment costs). The ideal treatment strategy of AR includes complete avoidance of allergens, local corticosteroids, leukotriene receptor antagonists, Th2 cytokine suppressors and nasal antihistamines, therapy. However, these therapeutic interventions show limited effectiveness and high cost of long-term treatment . Allergic rhinitis resistant to drug therapy usually submitted to posterior nasal nerve resection. This surgical maneuver was originated from Vidian neurectomy, which markedly reduces hypersecretion and hypersensitivity by ablation of the Vidian nerve with a transantral approach. However, Vidian neurectomy is occasionally accompanied by permanent comorbidities [e.g., reduced lacrimation and development of upper lip numbness Posterior nasal neurectomy is a novel alternative technique in which neural bundles - under direct vision- are selectively cut or cauterized at the sphenopalatine foramen. This enables avoidance of surgical compilations especially reduced lacrimation. However, literature is not yet addressed its safety and efficacy and no final consensus or guidelines had been drawn. In addition, it is of most importance to present our clinical experience and share our results regarding such procedure with the scientific community. The aim of this work was to present our clinical experience with endoscopic posterior nasal neurectomy in persistent allergic rhinitis.

Surgical technique: This procedure had been completed under general anesthesia. A 00 or a 300 nasal endoscope with a diameter of 4 mm is used throughout the surgery. About 1 mL of 1:100,000 epinephrine was injected at the posterior end of the middle meatus. Opening of the maxillary sinus and identification of its ostium to take it as a guide to reach the sphenopalatin foramen. Then in the middle meatus, a curved incision, 1.5cm long, had been made, starting from the superior margin of the inferior nasal turbinate up to the horizontal part of the ground lamella of the middle turbinate. The dissected mucosal flap had been separated from the vertical plate of the palatine bone, and the flap had been folded backwards until exposure of the sphenopalatine notch and the superior margin of the vertical plate of the palatine bone. Then, at the level of sphenopalatine foramen, the neurovascular bundle had been identified, with inclusion of the posterior nasal nerve. The PNN had identified and sectioned from the sphenopalatine artery only in four cases. The rest of cases, the whole bundle had been sectioned including the artery there is no significant side effects between both maneuvers. To avoid postoperative bleeding, a sufficient coagulation had been applied and nasal packing was inserted for 2 days

ELIGIBILITY:
Inclusion Criteria:

* Patients with allergic rhinitis
* Patients fit for surgery.

Exclusion Criteria:

* Coagulopathy, systemic diseases, and patients unfit for general anesthesia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-03-12 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
22-item Sino-Nasal Outcome Test (SNOT-22) | 6months after surgery
  each symptom is scored on a scale from 0 to 5 (0 = no problem, 1 = very mild problem, 2 = mild problem, 3 = moderate problem, 4 = severe problem and 5 = problem as bad as it can be).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Aouf, Principal Investigator — kafrelsheikh U
Locations (1):
- Kafrelsheikh university, Kafr ash Shaykh, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brozek JL, Bousquet J, Baena-Cagnani CE, Bonini S, Canonica GW, Casale TB, van Wijk RG, Ohta K, Zuberbier T, Schunemann HJ; Global Allergy and Asthma European Network; Grading of Recommendations Assessment, Development and Evaluation Working Group. Allergic Rhinitis and its Impact on Asthma (ARIA) guidelines: 2010 revision. J Allergy Clin Immunol. 2010 Sep;126(3):466-76. doi: 10.1016/j.jaci.2010.06.047. PMID 20816182
- [Background] Kobayashi T, Hyodo M, Nakamura K, Komobuchi H, Honda N. Resection of peripheral branches of the posterior nasal nerve compared to conventional posterior neurectomy in severe allergic rhinitis. Auris Nasus Larynx. 2012 Dec;39(6):593-6. doi: 10.1016/j.anl.2011.11.006. Epub 2012 Feb 15. PMID 22341334